CLINICAL TRIAL: NCT06239155
Title: Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of AST-3424 in Treatment of Patients With Advanced Solid Tumors and Its Correlation With AKR1C3 Enzyme Expression
Brief Title: A Phase I/II Study of AST-3424 in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascentawits Pharmaceuticals, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AST-3424-001
Record Dates: First submitted 2024-01-16; First posted 2024-02-02 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumors; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I: dose escalation phase (Experimental): AST-3424 (1.0 mg/m^2 to 10.0 mg/m^2 or higher doses) will be administered by IV infusion on Day1 and Day8 of each 21-day cycle. 1mg/m^2 and 2mg/m^2 cohort will enroll 1 participant respectively . 4mg/m^2 or higher dose cohorts will use 3+3 dose escalation design to determine the MTD and RP2D.
  Interventions: Drug: AST-3424
- Phase II: cohort expansion phase (Experimental): 6mg/m^2, administrated on Day1 and Day 8 of each 21-day cycle
  Interventions: Drug: AST-3424

INTERVENTIONS:
Drug: AST-3424 — liquid formulation for Intravenous infusion

SUMMARY:
An open-label, Phase I/II study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of AST-3424 administered as a single agent

DETAILED DESCRIPTION:
This is an open-label phase I/II clinical study to evaluate the safety, tolerability, MTD/RP2D, pharmacokinetics, preliminary efficacy, and the relationship between AKR1C3 expression and efficacy of AST-3424 monotherapy in advanced solid tumors.

The study is divided into phase I and Phase II. The maximum tolerated dose will be explored in phase I. In phase II, participants will be treated with AST-3424 according to the Phase I confirmed dose. Phase II clinical study will first be conducted in hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* phase I: dose escalation phase

  1. Male or female, 18-70 years old.
  2. Histologically and/or cytologically confirmed malignant solid tumors (including but not limited to hepatocellular carcinoma, intrahepatic cholangiocarcinoma, gastric cancer, esophageal cancer, colorectal cancer, pancreatic cancer, renal cell carcinoma, non-small cell lung cancer, and castration-resistant prostate cancer) that are metastatic or unresectable and have failed standard treatment or no standard treatment, pr not suitable for standard treatment at this stage.
  3. Once MTD is confirmed, participant in the Extended Dose group (MTD group) need to have at least one measurable lesion that meets the RECIST 1.1 criteria. Previously irradiated lesions are not measurable unless they show clear radiographic progression after radiotherapy.
  4. The physical status score of the Eastern Cancer Collaboration Group (ECOG) is 0 or 1.
  5. Life expectancy≥12 weeks.
  6. All toxicities (except alopecia, fatigue, or peripheral neuropathy) from previous anticancer therapy must have returned to grade 1 or baseline levels prior to initiation of the investigational drug (NCI CTCAE 5th Edition).
  7. The heart QTcF interval ≤450 ms in males or ≤ 470 ms in females.
  8. Laboratory tests must meet the following criteria. the indicators could not be corrected by blood transfusion or hematopoietic stimulating factors for 14 days prior to the screening laboratory examination.

     1. Hemoglobin ≥90 g/L
     2. Platelet count ≥100 x 10^9/L
     3. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
     4. Total bilirubin ≤ 1.5 x upper limit of normal(ULN)
     5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0× ULN, ≤ 5.0× ULN for liver tumors
     6. Creatinine clearance was > 50 mL/min according to Cockcroft-Gault formula
  9. No alcohol, drug or substance abuse history in the last 1 year.
  10. Fertile female patients should not breastfeeding and must have a negative pregnancy test result within 5 days before the start of treatment (positive urine pregnancy test result need to be confirmed by a serum pregnancy test)..
  11. Fertile female and male participant must consent to the use of an effective contraceptive method with their partner (e.g. surgical sterilization or condom or diaphragm contraception combined with spermicidal gel or intrauterine device (IUD), etc.) from the start of the study until 6 months after the last treatment.
  12. Voluntarily participate in this study, fully understand the relevant risks, have good compliance, and sign the informed consent.
* phase II: cohort expansion phase

  1. Male or female, ≥ 18 years old.
  2. Advanced HCC that is pathologically confirmed and cannot be controlled by surgical resection or local treatment.
  3. Prior treatment with standard systemic therapies, including but not limited to sorafenib and/or systemic chemotherapy containing oxaliplatin, lenvatinib, regorafenib and/or opdivo, disease progression, toxic intolerance or refusal to continue treatment with these drugs.
  4. At least one measurable lesion that meets RECIST 1.1 criteria. Lesions previously treated with radiotherapy are not measurable unless confirmed radiographic progression.
  5. Can provide pathological wax blocks or sections (including archived pathological wax blocks or sections) for AKR1C3 expression analysis, and be confirmed that AKR1C3 expression is strongly positive in liver tumor tissues (the proportion of tumor cells with AKR1C3 staining intensity of 2+ and/or 3+ is ≥70%, confirmed by the central laboratory using immunohistochemistry).
  6. The physical status score of the Eastern Cancer Collaboration Group (ECOG) is 0 or 1.
  7. Life expectancy≥12 weeks.
  8. With or without hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

     1. Participant with HBV infection must have HBV-DNA < 2,000 IU/ml and receive antiviral therapy with Entecavir, tenofovir disoproxil fumarate, and tenofovir alafenamide fumarate, according to National Guidelines for Chronic Hepatitis B Prevention and Treatment, maintained during the study period and continued until 6 months after the last dose.
     2. Participant with coexisting HCV infection (presence of detectable HCV-RNA or anti-HCV antibodies) can be treated according to medical practice.
  9. Child-Pugh score≤6.
  10. No history of hepatic encephalopathy.
  11. All toxicities (except alopecia, fatigue, or peripheral neuropathy) from previous anticancer therapy must have returned to grade 1 or baseline levels before initiating investigational drug use (NCI CTCAE 5th Edition).
  12. Laboratory tests must meet the following criteria. The indicators could not be corrected by blood transfusion or hematopoietic stimulating factors or albumin infusion within 14 days before the screening laboratory examination.

      1. Hemoglobin≥90 g/L
      2. Platelet count≥80 x 10^9/L
      3. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
      4. Serum total bilirubin ≤3 mg/dL
      5. ALT and AST ≤5.0 x ULN
      6. International Normalized Ratio (INR) ≤2.3 or prolonged prothrombin time ≤6 seconds
      7. Albumin≥29 g/L
      8. Creatinine clearance > 50 mL/min as measured by Cockcroft-Gault equation
  13. No alcohol, drug or substance abuse history in the last one year.
  14. Fertile female patients should not breastfeeding and must have a negative pregnancy test result within 5 days before the start of treatment (positive urine pregnancy test result need to be confirmed by a serum pregnancy test).
  15. Fertile female and male participant must consent to use effective contraceptive methods with their partner from the beginning of study participation (e.g., surgical sterilization or condom or diaphragm contraception combined with spermicidal gel or intrauterine device (IUD), etc.) until 6 months after the last treatment.

Voluntarily participate in this study, fully understand the risks involved, have good compliance, and sign informed consent. Participant may also sign a consent form for future biomedical research (FBR). However, participant who do not participate in the FBR may also participate in the principal trial.

Exclusion Criteria:

* phase I: dose escalation phase

  1. Untreated active central nervous system (CNS) metastases or leptomeningeal disease. Participant may participate in the study if their CNS metastases have been adequately treated and are stable for at least 4 weeks as confirmed by clinical examination and brain imaging (MRI or CT) during screening.
  2. Major surgery other than diagnostic surgery was performed within 4 weeks prior to initial dosing.
  3. Radiotherapy, surgery, chemotherapy, immunotherapy, cancer biotherapy, targeted therapy, or hormonal therapy within 4 weeks prior to the first dose (lomustine or mitomycin C treatment, requiring a 6-week washout period; Oral fluorouracil, requiring a 2-week washout period; Small molecule targeted therapy requires a 2-week washout period).
  4. Participated in an investigational drug (diagnostic or therapeutic) or device study within 4 weeks prior to initial dosing.
  5. Combined use of strong potent CYP3A4 inhibitors or inducers need to be used during the study.
  6. Uncontrolled, active bacterial, viral or fungal infections requiring systemic treatment.
  7. Known to be positive for human immunodeficiency virus (HIV) or syphilis.
  8. Women who are pregnant, breast-feeding, or planning to become pregnant.
  9. Concomitant diseases or symptoms that may interfere with the conduct of the study, or physical abnormalities that the investigator believes pose an excessive risk to the patient, including but not limited to active peptic ulcer or gastritis, changes in mental status, or mental abnormalities that may interfere with the patient's understanding of the informed consent form.
  10. Previous allergies to ethanol and propylene glycol.
  11. Unwilling or unable to comply with the study protocol for any reason.
* phase II: cohort expansion phase

  1. Untreated active central nervous system (CNS) metastases or leptomeningeal disease. Participant may participate in the study if their CNS metastases have been adequately treated and are stable for at least 4 weeks as confirmed by clinical examination and brain imaging (MRI or CT) during screening.
  2. A history of other malignancies within 2 years, except adequately treated basal cell carcinoma, carcinoma in situ at other sites, or other tumors whose natural history and treatment would not interfere with the evaluation of the safety and efficacy of the study.
  3. Major surgery other than diagnostic surgery was performed within 4 weeks prior to initial dosing.
  4. Radiotherapy, surgery, chemotherapy, immunotherapy, cancer biotherapy, targeted therapy, or hormonal therapy within 4 weeks prior to the first dose (lomustine or mitomycin C treatment, requiring a 6-week washout period; Oral fluorouracil, requiring a 2-week washout period; Small molecule targeted therapy requires a 2-week washout period).
  5. Participated in an investigational drug (diagnostic or therapeutic) or device study within 4 weeks prior to initial dosing.
  6. Combined use of strong potent CYP3A4 inhibitors or inducers need to be used during the study.
  7. Uncontrolled, active bacterial, viral or fungal infections requiring systemic treatment.
  8. Known active infection of human immunodeficiency virus (HIV) or syphilis.
  9. Clinically significant ascites，defined as those detected by physical examination and requiring control by abdominal puncture or additional pharmacological intervention to maintain symptoms (patients whose ascites detected only by imaging examination are eligible).
  10. Women who are pregnant, breast-feeding or planning to become pregnant.
  11. Concomitant diseases or symptoms that may interfere with the conduct of the study, or physical abnormalities that the investigator believes pose an excessive risk to the patient, including but not limited to history of gastrointestinal bleeding or high risk of bleeding within three months, active peptic ulcer or gastritis, changes in mental status, or mental abnormalities that may interfere with the patient's understanding of the informed consent form.
  12. Previous allergies to ethanol and propylene glycol.
  13. Unwilling or unable to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events(AEs) | measure begins from informed consent to 30 days after last dose of study drug.
  Adverse events will be noted and graded according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0 or severity (if not covered by CTCAE)
Safety changes in electrocardiogram (ECG) | Day 1 Cycles 1 and 2 (each cycle is 21 days)
  Resting 12-lead ECGs will be obtained from all subjects' pre-AST-3424 infusion and within 30 minutes post-AST-3424 infusion in order to assess any impact AST-3424 may have on the QT interval as assessed by the Fridericia's Correction Formula (QTcF).
Safety Changes of body weight | Day 1 of each cycle (there are 34 cycles; 21 days for each cycle)
  If during treatment a participant's body weight changes by >10%, the dose should be adjusted.
Dose limiting toxicities (DLTs) in phase I | Throughout Cycle 1 (21 days for each cycle) in phase I (dose escalation phase).
  Number of participants with dose limiting toxicities (DLTs)
Maximum Tolerated Dose(MTD)/Recommended Phase 2 Dose (RP2D) in phase I | Day 1 and Day 8 of each cycle (all 34 cycles and there are 21 days for each cycle)
  Determination of the MTD, based on the frequently of DLTs observed in Cycle 1 in participants enrolled to the Dose Escalation Phase.
Pharmacokinetics (PK) - Time to maximum concentration (Tmax) | Days 1 and 8 of Cycle 1 (first cycle of 34 cycles and there are 21 days for each cycle)
  Tmax of AST-3424 and AST-2660 will be computed for each subject where possible.
PK - Maximum peak plasma concentration (Cmax) | Days 1 and 8 of Cycle 1 (first cycle of 34 cycles and there are 21 days for each cycle)
  Cmax of AST-3424 and AST-2660 will be computed for each subject where possible.
PK - The magnitude of the slope of the linear regression of the log concentration vs. time profile during the terminal phase (Kel) | Days 1 and 8 of Cycle 1 (first cycle of 34 cycles and there are 21 days for each cycle)
  Kel of AST-3424 and AST-2660 will be computed for each subject where possible.
PK - Half-life (T1/2) | Days 1 and 8 of Cycle 1 (first cycle of 34 cycles and there are 21 days for each cycle)
  T1/2 computed as ln (2)/Kel of AST-3424 and AST-2660 will be computed for each subject where possible.
PK - Area under the concentration-time curve (AUClast) | Days 1 and 8 of Cycle 1(first cycle of 34 cycles and there are 21 days for each cycle)
  AUClast from Hour 0 through the last quantifiable concentration time (LQCT), where LQCT is the time at which the last sample with a quantifiable concentration was drawn
Objective response rate(ORR) | Approximately 36 months
Disease control rate(DCR) | Approximately 36 months
Duration of response (DOR) | Approximately 36 months
Progress free survival (PFS) | Approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai East Hospital; Shukui Qin, Principal Investigator — Chinese People's Liberation Army Eastern Theater General Hospital Qinhuai medical District
Locations (7):
- China (7):
  - Guangdong Qifu Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Chinese People's Liberation Army Eastern Theater General Hospital Qinhuai medical District, Nanjing, Jiangsu
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided